CLINICAL TRIAL: NCT07016984
Title: Effect of Light Intensity Reduction During Mydriasis on the Comfort Level in Premature Infants Undergoing Retinopathy of Prematurity Screening
Brief Title: Comfort Level in Premature Infants Undergoing Retinopathy of Prematurity Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Alev Sivasli, Principal Investigator, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Decision No:2023/44
Record Dates: First submitted 2025-05-29; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Premature; Retinopathy of Prematurity; Pain
Keywords: infant comfort; Light Exposure; Mydriasis; Non-pharmacological intervention; Neonatal intensive care; Premature infants; Retinopathy of prematurity
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity; Pain; Mydriasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): Following the mydriasis procedure performed prior to ROP examination, the eyes were covered with these patches.
  Interventions: Other: standard phototherapy eye patches
- Control Group (No Intervention): During the ROP examination, no eye patching was applied.

INTERVENTIONS:
Other: standard phototherapy eye patches — Following the mydriasis procedure performed prior to ROP examination, the eyes were covered with these patches.
  Arms: Experimental Group

SUMMARY:
Retinopathy of prematurity (ROP) screening is a routine yet painful procedure for premature infants, often necessitating pharmacological mydriasis. The associated light exposure due to dilated pupils can increase stress and reduce infant comfort. This study aimed to investigate the effect of using a phototherapy eye mask during mydriasis on the comfort levels of premature infants.

DETAILED DESCRIPTION:
Retinopathy of prematurity is a pathological condition affecting the developing retinal blood vessels in low birth weight premature infants and is one of the leading causes of childhood blindness. In recent years, advancements in neonatal intensive care in developing countries such as China, India, and Turkey have increased the survival rates of premature infants, consequently raising the number of infants requiring ROP screening examinations. Health Organization (WHO) recommends conducting the initial ROP examination before the infant is discharged from the hospital. However, ROP screening is a painful and stressful procedure that includes the administration of mydriatic agents, the insertion of a speculum to open the palpebral fissure, and scleral depression to visualize the retinal periphery. These interventions often result in discomfort and distress for the infant. Globally, most newborns admitted to neonatal intensive care units (NICUs) undergo repeated painful procedures. It is well-established that premature infants can perceive pain, and exposure to pain during the early stages of life may lead to long-term neurological consequences. In very preterm infants, early exposure to procedural pain has been associated with impaired cognitive development and reductions in frontal and parietal lobe volumes, brain size, white matter, and subcortical gray matter. Considering the frequency of painful interventions during hospitalization, gaining deeper insight into stress-inducing factors and exploring methods to enhance infant comfort is of great importance. Various non-pharmacological interventions-such as pacifiers, music, and oral sucrose-have been studied for their effectiveness in reducing pain and stress during ROP examinations. However, research evaluating the effect of minimizing light exposure during pupil dilation (mydriasis) is limited. Mydriatic eye drops, used to dilate the pupils for examination, are known to cause light sensitivity and photophobia. It is hypothesized that the increased light sensitivity resulting from pupil dilation before the examination contributes to infant discomfort and stress. Therefore, this study aims to investigate the effect of reducing light exposure-by applying eye patches during the mydriasis process-on the comfort levels of premature infants undergoing ROP screening.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤34 weeks
* Birth weight ≤1700 grams
* Parental consent to participate in the study

Exclusion Criteria:

* Required mechanical ventilation during the study period
* Had genetic disorders, heart disease, neurological or metabolic conditions, pulmonary anomalies, or ocular malformations
* Had any conditions affecting the stress response
* Were administered sedatives, muscle relaxants, corticosteroids, or analgesics
* Had major congenital anomalies

Min Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
post-test total and subdimension scores from the Premature Infant Comfort Scale (PICS), along with the statistical comparisons between the two groups | 8 hours
  Statistically significant differences were observed in the total scores and all subdimensions of the PICS-alertness, calmness/agitation, crying (in non-ventilated infants), physical movement, muscle tone, facial movements, and average heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin Cigdem, Associate Professor, Study Director — Topkapi University, Istanbul, Turkey; Nurşah B Şamlıer, PhD, Principal Investigator — Nisantasi University, Istanbul, Turkey
Locations (1):
- Nisantasi University, Sarıyer, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
They are fully familiar with the study in all its details, so I do not find it necessary to elaborate further in order to avoid wasting time.